CLINICAL TRIAL: NCT04754347
Title: Randomized, Controlled Trial of a Computer Aided Detection Device in Standard Colonoscopy
Brief Title: Computer Aided Detection of Polyps in Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iterative Scopes, Inc (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Pro00047634
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Polyp
Keywords: Screening Colonoscopy; Artificial Intelligence; Computer Aided Detection; Adenoma Detection Rate; Adenomas per Colonoscopy; Surveillance Colonoscopy; Colorectal Cancer; Software as a Medical Device
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Routine Colonoscopy
- Experimental (Experimental): Routine Colonoscopy with the use of Skout
  Interventions: Device: Computer Aided Detection device

INTERVENTIONS:
Device: Computer Aided Detection device — The Computer Aided Detection device, Skout, is designed to help endoscopists detect potential colorectal polyps during colonoscopies. The system performs automated real-time analysis on endoscopic video data to identify potential polyps and produces an informational visual aid around the appropriate sections of the video frames on a display monitor.
  Arms: Experimental

SUMMARY:
The aim of this study is to evaluate the clinical benefit and safety of using a computer aided detection device, Skout, for real-time polyp detection in colonoscopy procedures with the indication of screening or surveillance. One of the reasons for the development of interval colorectal cancers is polyps missed during colonoscopy. Our hypothesis is that with the aid of Skout, the adenomas detected per colonoscopy will increase, and it is plausible to believe that this increase in detection could reduce the incidence of interval cancers.

ELIGIBILITY:
Inclusion Criteria

Participants will be eligible for this study if they are:

* Undergoing colonoscopy with screening, surveillance, or diagnostic indications.
* Undergoing a procedure by a participating endoscopist.
* Have given informed consent.

Exclusion Criteria

Participants will not be eligible for this study if they:

* Have a history of inflammatory bowel disease.
* Have a history of familial adenomatous polyposis.
* Are under the age of 40.
* Have had a colonoscopy within the previous three (3) years.
* Undergoing diagnostic colonoscopy with high-risk indications including iron deficiency anemia, abnormal CT imaging, unexplained weight loss, Lynch Syndrome, blood in stool or FIT positive test.
* Entered with poor bowel preparation (inadequate for procedure as assessed by the Investigator).
* Use anti-platelet agents or anticoagulants that preclude the removal of polyps during the procedure.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1472 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Adenomas per colonoscopy | At the end of the procedure, 1 day
  The total number of adenomas detected divided by the total number of colonoscopies.
Positive predictive value | At the end of the procedure, 1 day
  The total number of adenomas and serrated lesions detected divided by the total number of extractions.

SECONDARY OUTCOMES:
Adenoma detection rate | At the end of the procedure, 1 day
  The percentage of participants aged ≥50 years undergoing first-time screening colonoscopy who have one or more conventional adenomas detected.
Sessile serrated lesions detected | At the end of the procedure, 1 day
  The total number of polyps with histology or serrated adenoma, traditional serrated adenoma or serrated lesion with cytological dysplasia, excluding hyperplastic polyps.
Colorectal cancer surveillance interval | At the end of the procedure, 1 day
  The mean recommended timeframe for follow up colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Aasma Shaukat, MD, MPH, Principal Investigator — University of Minnesota
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mount Auburn Hospital, Cambridge, Massachusetts
  - MNGI Digestive Health, Plymouth, Minnesota
  - Concord Endoscopy Center, Concord, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaukat A, Lichtenstein DR, Somers SC, Chung DC, Perdue DG, Gopal M, Colucci DR, Phillips SA, Marka NA, Church TR, Brugge WR; SKOUT Registration Study Team. Computer-Aided Detection Improves Adenomas per Colonoscopy for Screening and Surveillance Colonoscopy: A Randomized Trial. Gastroenterology. 2022 Sep;163(3):732-741. doi: 10.1053/j.gastro.2022.05.028. Epub 2022 May 25. PMID 35643173